CLINICAL TRIAL: NCT01928186
Title: Imaging Early Response of ER+, HER2- Breast Cancer to Aromatase Inhibitor (AI) +/- Ovarian Suppression (OS) Therapy With [18F]Fluorothymidine (FLT) PET
Brief Title: FLT PET in Measuring Treatment Response in Patients With Newly Diagnosed Estrogen Receptor-Positive, HER2-Negative Stage I-III Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Hannah Linden, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 7536; NCI-2013-01380 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 7536 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH); RC1CA146456 (NIH)
Record Dates: First submitted 2013-08-20; First posted 2013-08-23 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-04

CONDITIONS: Estrogen Receptor Positive; HER2/Neu Negative; Male Breast Carcinoma; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — alovudine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic (FLT PET) (Experimental): Patients undergo FLT PET at baseline and 1-6 weeks after the start of treatment.
  Interventions: Drug: Fluorothymidine F-18; Procedure: Positron Emission Tomography; Other: Laboratory Biomarker Analysis; Drug: Run-in (short pre-surgery course) of endocrine-targeted therapy

INTERVENTIONS:
Drug: Fluorothymidine F-18 — Undergo FLT PET
  Other Names: 18F-FLT; 3'-deoxy-3'-[18F]fluorothymidine
Procedure: Positron Emission Tomography — Undergo FLT PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Run-in (short pre-surgery course) of endocrine-targeted therapy — Patients undergo run-in (short pre-surgery course) of endocrine-targeted therapy with aromatase inhibitor between the two (baseline and repeat) FLT PET scans. This is not an experimental therapy. This is a standard of care therapy that patients will continue after surgery, when the study is completed.

SUMMARY:
This clinical trial studies fluorine F 18 fluorothymidine (FLT) positron emission tomography (PET) in measuring treatment response in patients with newly diagnosed estrogen receptor (ER)-positive, human epidermal growth factor receptor 2 (HER2)-negative stage I-III breast cancer. Comparing results of diagnostic procedures done before and during hormone therapy may help doctors predict a patient's response to treatment and help plan the best treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Measure the effect of a short course of endocrine therapy on primary breast cancer metabolism and proliferation by measuring changes in serial FLT PET measures pre and post a short course of endocrine therapy.

SECONDARY OBJECTIVES:

I. Compare changes in imaging measures to tissue measures of response, in particular antigen identified by proliferation-related Ki-67 antigen (Ki-67), in the pre-therapy biopsy versus the post-therapy surgical specimen.

II. Correlate imaging measures to measures of gene expression from pre and post therapy assays to determine if there are molecular changes associated with early response to therapy.

OUTLINE:

Patients undergo FLT PET at baseline and 1-6 weeks after the start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* A new diagnosis of invasive breast cancer > 1.0 cm in size, ER+ clinical stage I-III
* Patient must have surgical resection followed by systemic adjuvant therapy with an aromatase inhibitor (AIs) as part of planned treatment; any approved AI at standard clinical dosing may be used; in pre-menopausal patients, ovarian suppression with a gonadotropin-releasing hormone (GnRH) agonist will be started prior to initiation of the AI on a separate clinical trial in parallel with the imaging study
* Have tissue block available from core biopsy for correlative biomarkers and genomic assay
* Have menopausal status determined prior to study enrollment; for study purposes, postmenopausal is defined as

  * A prior documented bilateral oophorectomy, or
  * A history of at least 12 months without spontaneous menstrual bleeding, or
  * Age 60 or older with a prior hysterectomy without oophorectomy, or
  * Age less than 60 with a prior hysterectomy without oophorectomy (or in whom the status of the ovaries is unknown) with a documented follicle-stimulating hormone (FSH) level demonstrating confirmatory elevation in the postmenopausal range for the lab
* Negative pregnancy test within 7 days of baseline positron emission tomography (PET) scan for pre-menopausal patients
* Tumor HER2/neu expression must be determined (as part of standard clinical care) prior to study enrollment; HER2 may be tested by any Food and Drug Administration (FDA) approved HER2 testing method; if determination is intermediate by immunohistochemistry (IHC), fluorescent in situ hybridization (FISH) or another alternate HER2 test must be performed
* Be a candidate for [18F]FLT PET imaging
* Be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific screening procedures
* Be willing and able to comply with scheduled visits and other trial procedures

Exclusion Criteria:

* Current use of aromatase inhibitor as prevention or treatment for breast cancer
* Life expectancy of less than two months
* HER2/neu positive by IHC and/or another FDA approved HER2 testing method
* Inability to tolerate scanning (e.g. - claustrophobia, severe pain)
* Weight exceeding capacity of imaging table

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-09; Primary Completion 2015-07-20 (Actual); Study Completion 2015-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Linden, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (FLT PET)
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Diagnostic (FLT PET): Patients with early stage, ER positive primary breast cancer undergo FLT PET scan at baseline and 1-6 weeks after the start of standard endocrine treatment. The surgery follows 1-7 days after the second FLT PET scan.
  Tracer used in the FLT PET (positron emission tomography) scanning procedure: [F18] fluorothymidine.
  Positron Emission Tomography: Undergo FLT PET
  Laboratory Biomarker Analysis: Correlative studies - Ki67 staining of the tumor tissue in the biopsy and surgical specimen.
Arm/Group | Diagnostic (FLT PET)
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 60.4 [28.2 to 74.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Clinical stage [Count of Participants; unit: Participants] — Patients presented in early clinical stages of breast cancer, with the extent of disease increasing from the stage I to IIB, as indicated in the NCI TNM staging system (v. 07/11/2014):
  Stage I: T1 N0; Stage IIA: T0 N1 or T1 N1 or T2 N0; Stage IIB: T2 N1 or T3 N0. Definitions: No evidence of primary tumor (T0); Primary tumor < or = 20 mm (T1); Primary tumor >20 mm but < or = 50 mm (T2); Primary tumor > 50 mm (T3); No regional lymph node metastases (N0); Metastases to movable ipsilateral level I, II axillary lymph nodes (N1).
  Participants
    Stage I | 10
    Stage IIA | 14
    Stage IIB | 4

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Net Influx Constant (Ki) by FLT PET
Description: Percent change between pre-treatment (baseline) and post-therapy PET measurements in breast tumors will be computed.
  Association between Ki-67 and Ki by FLT (KFLT) decline will be analyzed using the mid-P adjustment to Fisher's exact test to evaluate the potential clinical utility of change in FLT as a biomarker for early response, using Ki-67 as the standard for early response.
Time Frame: Baseline to up to 6 weeks
Measure: Median (Full Range); unit: % change
Arm/Group | Diagnostic (FLT PET)
Number analyzed (Participants) | 28
% change | -32.0 [-82.4 to 3953.7]
Statistical Analysis 1: Comparison: Diagnostic (FLT PET); Association between response assessed by Ki-67 protein staining (i.e. < 10% positive cells in the surgical sample) and by the influx constant Ki decline (i.e. 30 % or larger decline between the baseline and post-therapy FLT PET) was analyzed using the mid-P adjustment to Fisher's exact test; Test type: Other; p = 0.51, Fisher Exact; the mid-P adjustment to Fisher's exact test

2. Primary Outcome: Percent Change in SUV by FLT PET
Description: Percent change between pre-treatment (baseline) and post-therapy measurements of FLT standardized uptake value (SUV) in breast tumors will be computed.
Time Frame: Baseline to up to 6 weeks
Measure: Median (Full Range); unit: % change
Arm/Group | Diagnostic (FLT PET)
Number analyzed (Participants) | 28
% change | -26.6 [-77.3 to 7.4]

3. Primary Outcome: Percentage of Ki-67 Positive Tumor Cells in Surgical (Post-therapy) Sample
Description: Surgically removed breast tumor tissue is stained using immuno-histochemistry techniques to visualize dividing cells expressing the Ki-67 protein, which is a cellular marker for proliferation.
Time Frame: 1 to 6 weeks post-therapy start
Measure: Median (Full Range); unit: % stained cells
Arm/Group | Diagnostic (FLT PET)
Number analyzed (Participants) | 28
% stained cells | 3 [0 to 40]

4. Primary Outcome: Percentage Change in Ki-67 Positive Cells Between Pre-therapy and Post-therapy Tumor Specimens
Description: Tumor tissue samples from pre-treatment (baseline) biopsy and post-treatment surgery are stained using immuno-histochemistry techniques to visualize dividing cells expressing the Ki-67 protein, which is a cellular marker for proliferation.
  The % values of positive cells from the baseline and post-treatment samples are then compared for each individual patient.
  Association between Ki-67 and KFLT decline will be analyzed to evaluate the potential clinical utility of change in FLT as a biomarker for early response, using Ki-67 as the standard for early response.
Time Frame: Baseline to up to 6 weeks
Measure: Median (Full Range); unit: % change
Arm/Group | Diagnostic (FLT PET)
Number analyzed (Participants) | 28
% change | -80.0 [-100.0 to 400.0]

5. Secondary Outcome: Percentage Change in K1 (Blood Flow Parameter) by FLT PET
Description: Percent change between pre-treatment (baseline) and post-therapy PET measurements in breast tumors will be computed.
Time Frame: Baseline to up to 6 weeks
Measure: Median (Full Range); unit: % change
Arm/Group | Diagnostic (FLT PET)
Number analyzed (Participants) | 28
% change | -6.2 [-94.6 to 262.1]

6. Secondary Outcome: Baseline Ki (Flux Constant) Values by FLT PET
Description: Ki (flux constant) in breast tumor tissue as determined by the pre-therapy (baseline) FLT PET scan
Time Frame: Baseline
Measure: Median (Full Range); unit: mL/min/mL
Arm/Group | Diagnostic (FLT PET)
Number analyzed (Participants) | 28
mL/min/mL | 0.015 [0.0025 to 0.0353]

7. Secondary Outcome: Baseline FLT Transport (K1) Values by FLT PET
Description: K1 (blood flow measure) in breast tumor tissue as determined by the pre-therapy (baseline) FLT PET
Time Frame: Baseline
Measure: Median (Full Range); unit: mL/min/mL
Arm/Group | Diagnostic (FLT PET)
Number analyzed (Participants) | 28
mL/min/mL | 0.0501 [0.0119 to 0.3699]

8. Secondary Outcome: Baseline Standardized Uptake Values (SUV) by FLT PET
Description: FLT SUV in breast tumor tissue as determined by the pre-therapy (baseline) FLT PET
Time Frame: Baseline
Measure: Median (Full Range); unit: g/mL
Arm/Group | Diagnostic (FLT PET)
Number analyzed (Participants) | 28
g/mL | 2.5 [1.06 to 7.77]

9. Secondary Outcome: Post-therapy Ki (Flux Constant) Values by FLT PET
Description: Ki (flux constant) in breast tumor tissue as determined by the post-therapy FLT PET
Time Frame: 1 to 6 weeks post-therapy start
Measure: Median (Full Range); unit: mL/min/mL
Arm/Group | Diagnostic (FLT PET)
Number analyzed (Participants) | 28
mL/min/mL | 0.0142 [0.0015 to 0.0352]

10. Secondary Outcome: Post-treatment FLT Transport (K1) Values by FLT PET
Description: K1 (blood flow measure) in breast tumor tissue as determined by the post-therapy FLT PET
Time Frame: 1 to 6 weeks post-therapy start
Measure: Median (Full Range); unit: mL/min/mL
Arm/Group | Diagnostic (FLT PET)
Number analyzed (Participants) | 28
mL/min/mL | 0.0675 [0.0018 to 0.4335]

11. Secondary Outcome: Post-treatment Standardized Uptake Values (SUV) by FLT PET
Description: FLT SUV in breast tumor tissue as determined by the post-treatment FLT PET
Time Frame: 1 to 6 weeks post-therapy start
Measure: Median (Full Range); unit: g/mL
Arm/Group | Diagnostic (FLT PET)
Number analyzed (Participants) | 28
g/mL | 1.76 [0.76 to 3.78]

12. Other Pre Specified Outcome: Post-treatment Gene Expression Levels
Description: Analyzed using BeadStudio software. Four clustering metrics for calculating dissimilarities (correlation, absolute correlation, Euclidean, and Manhattan) are available in BeadStudio and will be applied using standard analysis methods and diagnostics in BioConductor. To focus the analysis, proposed gene sets will be examined based on biological pathways and molecular signatures.
Time Frame: 1 to 6 weeks post-therapy start
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Pre-treatment Gene Expression Levels
Description: as for outcome 12
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Diagnostic (FLT PET)
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 1/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (FLT PET) (N=28)
Infiltration at injection site (Injury, poisoning and procedural complications) | 1 (1) — Infiltration at injection site detected on imaging, without clinical symptoms

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No